CLINICAL TRIAL: NCT01573845
Title: The GREEN (Growing Right: Eating Eco-Friendly & Nutritious) Project Lunch Box Study
Brief Title: The GREEN Project Lunch Box Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R01HD065888-01 (NIH); 1R01HD065888 (NIH)
Record Dates: First submitted 2012-04-03; First posted 2012-04-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Health Communication
Keywords: child; communication; diet; food; health communication; nutrition; parents; primary schools; school age population; school health
MeSH Terms: conditions — Communication | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Eating + Eco-Friendly Campaign (Experimental)
  Interventions: Behavioral: Healthy Eating + Eco-Friendly Campaign
- Healthy Eating Campaign (Active Comparator)
  Interventions: Behavioral: Healthy Eating Campaign
- Control/Delayed Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Healthy Eating + Eco-Friendly Campaign — Participants receive a 6-month school-based campaign that includes:
  * A 22-lesson classroom curriculum
  * Homework activities that involve the family
  * Monthly parent newsletters
  * A food shopping and packing guide for parents
  * Food demonstrations
  * A poster contest
  * School wide announcements
  Arms: Healthy Eating + Eco-Friendly Campaign
Behavioral: Healthy Eating Campaign — Participants receive a 6-month school-based campaign that includes:
  * A 22-lesson classroom curriculum
  * Homework activities that involve the family
  * Monthly parent newsletters
  * A food shopping and packing guide for parents
  * Food demonstrations
  * A poster contest
  * School wide announcements
  Arms: Healthy Eating Campaign

SUMMARY:
The central hypothesis of The GREEN Project Lunch Box Study is that a school-based communication campaign that combines healthy eating and eco-friendly messages will improve the quality of foods that children bring from home to school more than a healthy eating campaign alone and compared to a control/delayed intervention condition at the end of one school year.

DETAILED DESCRIPTION:
The proposed intervention seeks to improve the quality of foods brought to school from home by taking advantage of a natural synergy between healthy eating and eco-friendly behaviors to increase motivation to adopt healthy eating behaviors. The project involves the design, implementation and evaluation of a novel, school based communications campaign to simultaneously improve the nutrition quality and eco-friendliness of foods that elementary school children bring from home to school.

The intervention is a theory-based multi-channel communications campaign based on qualitative research with the target population: children in grades three and four in public schools in Eastern Massachusetts and their caregivers. Schools were randomized to one of three conditions: (1) a campaign that includes healthy eating and eco-friendly messages; (2) a campaign that includes healthy eating messages only; and (3) a delayed healthy eating eco-friendly campaign after serving as a control group. Foods brought from home and the packaging associated with those foods will be assessed at baseline and at the end of the school year using a photographic technique.

The primary outcome of interest is change in the number of servings of fruits and vegetables. Secondary outcomes will include changes in the quantity of sugar-sweetened beverages; changes in processed, energy-dense foods; and changes in sugar sweetened beverages brought from home. We will also be able to assess changes in trash associated with foods brought from home.

ELIGIBILITY:
CHILD PARTICIPANTS

Inclusion Criteria:

* 3rd or 4th grade student in participating classroom
* Brings food from home to school at least 3 days per week

Exclusion Criteria:

* Not a 3rd or 4th grade student
* Not enrolled in a participating classroom
* Does not bring food from home to school at least three days per week

PARENT/CARETAKER PARTICIPANTS

Inclusion Criteria:

* Child is a 3rd or 4th grade student in participating classroom
* Child brings food from home to school at least 3 days per week

Exclusion Criteria:

* Child is not a 3rd or 4th grade student
* Child is not enrolled in a participating classroom
* Child does not bring food from home to school at least three days per week

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Changes in the quantity of fruit and vegetables brought from home to school | 6 months

SECONDARY OUTCOMES:
Changes in the quantity of sugar-sweetened beverages brought from home to school | 6 months
Changes in the quantity of processed, energy-dense foods brought from home to school | 6 months
Changes in trash weight associated with foods brought from home to school | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne P Goldberg, PhD, RD, Principal Investigator — Tufts University

REFERENCES:
- [Result] Hubbard KL, Must A, Eliasziw M, Folta SC, Goldberg J. What's in children's backpacks: foods brought from home. J Acad Nutr Diet. 2014 Sep;114(9):1424-31. doi: 10.1016/j.jand.2014.05.010. Epub 2014 Jul 16. PMID 25037557
- [Result] Goldberg JP, Folta SC, Eliasziw M, Koch-Weser S, Economos CD, Hubbard KL, Tanskey LA, Wright CM, Must A. Great Taste, Less Waste: a cluster-randomized trial using a communications campaign to improve the quality of foods brought from home to school by elementary school children. Prev Med. 2015 May;74:103-10. doi: 10.1016/j.ypmed.2015.02.010. Epub 2015 Feb 28. PMID 25735605